CLINICAL TRIAL: NCT05791617
Title: PET/MR in Post Stroke Cardiac Inflammation Study
Acronym: PEPSI
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-22-507
Record Dates: First submitted 2023-02-08; First posted 2023-03-30 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Inflammation
Keywords: stroke; PET/MRI; Inflammation; Heart
MeSH Terms: conditions — Stroke; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (Ischemic stroke): Left and right middle cerebral artery ischemic stroke Patients presenting with acute onset focal neurological deficits and DWI-MRI evidence of an acute brain infarct of the left or right middle cerebral artery ischemic stroke.
  Interventions: Diagnostic Test: cardiac PET/MRI; Diagnostic Test: Inflammatory markers; Diagnostic Test: Diagnostic Test: NT-proBNP
- Controls (TIA): Patients with acute focal neurological symptoms without brain infarct on MRI. Patients presenting with acute onset focal neurological deficits presumed to be of vascular origin, WITHOUT DWI-MRI evidence of an acute brain infarct.
  Interventions: Diagnostic Test: cardiac PET/MRI; Diagnostic Test: Inflammatory markers; Diagnostic Test: Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: cardiac PET/MRI — Patients will undergo cardiac PET/MRI scanning at 30±5 days and at 90±5 days post-stroke.
Diagnostic Test: Inflammatory markers — Measurement of a panel of 92 systemic inflammatory markers on patients' blood samples at 30±5 days and at 90±5 days post-stroke
  Other Names: Olink® Target-96 inflammatory biomarker panel
Diagnostic Test: Diagnostic Test: NT-proBNP — NT-proBNP is useful both in the diagnosis and prognosis of heart failure and is considered to be a gold standard biomarker in heart failure. Measurement of NT-proBNP on patients' blood samples at 30±5 days and at 90±5 days post-stroke
  Other Names: N-terminal prohormone of brain natriuretic peptide

SUMMARY:
Patients with stroke have a 25x higher risk of cardiovascular complications within the first 30 days of the event compared to individuals without stroke. The mechanisms behind these complications are not well understood. Evidence suggests that inflammation plays a central role. With the present proof-of-concept prospective cohort study, the investigators aim to demonstrate that patients develop cardiac inflammation after stroke by performing positron emission tomography (PET) magnetic resonance imaging (MRI) of the heart within 15 days after stroke. As a secondary aim, the investigators will evaluate whether post-stroke cardiac inflammation persists at 3 months after stroke. The control group will be comprised of age- and sex-matched individuals without stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years willing to cons Age ≥18 years willing to consent
* Patients with acute ischemic stroke in the right or left MCA territory, admitted to University Hospital, London Health Sciences Centre (LHSC) or evaluated at LHSC's Urgent TIA and Stroke Prevention Clinic. Acute ischemic stroke is defined as acute onset focal symptoms matching an acute brain infarct documented on a Head CT or on diffusion weighted imaging (DWI) MRI of the brain showing restricted diffusion.
* Willing to consent.

Exclusion Criteria:

* History of known heart disease defined as known atrial fibrillation, prior myocardial infarction, coronary artery disease, heart failure, prior cardiovascular surgery or percutaneous intervention
* Stroke in the previous 3 months before the qualifying stroke.
* High-sensitivity Troponin-T (HS-TnT) >100 ng/L on routine standard of care acute stroke bloodwork.
* Clinically or neurologically unstable patients as per the treating physician.
* Ongoing infection or recent infection within the previous 3 months.
* Surgery within 3 months before the stroke.
* Concurrent inflammatory conditions (connective tissue diseases, rheumatological disease, etc.) or use of anti-inflammatory medications.
* Contraindications to the use of gadolinium (e.g., pregnancy, stage IV renal insufficiency)
* Subjects will be excluded if they fail the St. Joseph's Health Care standard MRI screening questionnaire. Briefly, this questionnaire screens for: Heart Pacemakers / Wires, Aneurysm Clips, Shunt / Surgical Clips, Shrapnel / Bullets, Dentures or Metal braces, Intra-Uterine Device, Heart Valves, Ear Implants, Prostheses, Medication Patches (Nicoderm, Habitrol, Transderm-Nitro, etc.), Claustrophobia, History of a head or eye injury involving metal fragments. Patients with an eGFR < 40 will be excluded, as impaired renal function places the patient at a higher risk for a rare reaction to Gd-DTPA, the MRI contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise 4 patients with acute ischemic stroke in the right MCA territory involving the insular cortex, 4 patients in the left MCA territory involving the insular cortex, and 4 age- and sex-matched individuals presenting with acute stroke symptoms but no evidence of stroke on brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Cardiac Inflammation Levels at 30±5 Days Post-Stroke measured by PET/MR Scanning | At 30 days±5 post stroke
  Cardiac inflammation as measure on PET/MR scanning.
Cardiac Inflammation Levels at 90±5 Days Post-Stroke measured by PET/MR Scanning | At 90±5 days compared to first 30 days±5 post-stroke
  Cardiac inflammation as measure on PET/MR scanning.

SECONDARY OUTCOMES:
Change in B-Type Natriuretic Peptide (NT-proBNP) and HS-TnT levels between 30±5 days and 90±5 days post-stroke. | At 90±5 days compared to first 30±5 days post stroke
  Change in levels of NT-proBNP and HS-TnT between 30±5 and 90±15 days post-stroke.
Change in systemic inflammatory markers between 30±5 and 90±5 days post-stroke | At 90±5 days compared to first 30±5 days
  Systemic inflammatory markers will be measured using a high-performance biomarker panel for the following 92 proteins (all of which will be informed in pg/mL):
  ADA; ARTN; AXIN1; NGF; CCL13; CCL19; CCL2; CCL20; CCL23; CCL25; CCL28; CCL3; CCL4; CCL7; CCL8; CXCL10; CXCL11; CXCL5; CXCL6; CXCL9; CDCP1; CASP8; CST5; DNER; CCL11; EIF4EBP1; FGF19; FGF21; FGF23; FGF5; FLT3LG; CX3CL1; GDNF; CXCL1; HGF; IFNG; IL1A; IL10; IL10RA; IL10RB; IL12B; IL13; IL15RA; IL17A; IL17C; IL18; IL18R1; IL2; IL2RB; IL20; IL20RA; IL22RA1; IL24; IL33; IL4; IL5; IL6; IL7; CXCL8; MMP1; KITLG; LIF; LIFR; LTA; CSF1; SIRT2; CD244;NTF3;NRTN;OSM;CD274;S100A12;TGFA;STAMBP;SLAMF1;MMP10;SULT1A1;CD6;CD5;CD8A;TSLP;TGFB1;TNF;TNFSF10;TNFSF11;TNFSF12;TNFSF14;TNFRSF11B;CD40;TNFRSF9;PLAU;VEGFA

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Sposato, MD, Principal Investigator — London Health Sciences Center, Western University
Locations (1):
- Heart & Brain Lab, Western University, London, Ontario, Canada